CLINICAL TRIAL: NCT00779532
Title: A Randomized, Double-blind, Placebo and Positive Controlled, Parallel Group Trial to Investigate the Effect of Multiple Doses of NOMAC-E2 on QT/QTc Interval in Healthy Women
Brief Title: Thorough QT/QTc Study of Multiple Oral Doses of NOMAC-E2 (Org 10486 0 + Org 2317) in Healthy Women (Study 292011)(P05802)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: P05802; EudraCT # 2008-001649-25; 292011
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Contraception
Keywords: Electrocardiography; Pharmacokinetics
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Active Comparator): Once daily intake (orally) of 5 NOMAC-E2 placebo tablets from Day -1 to Day 14.
  Once daily intake (orally) of one moxifloxacin placebo capsule at Day -1.
  Once daily intake (orally) of one moxifloxacin capsule of 400 mg at Day 14.
  Interventions: Drug: Moxifloxacin; Drug: Moxifloxacin placebo; Drug: NOMAC-E2 placebo
- Group B (Experimental): Once daily intake (orally) of 4 NOMAC-E2 placebo tablets and 1 NOMAC-E2 (2.5/1.5 mg) tablet from Day 1 to Day 14.
  Once daily intake (orally) of 5 NOMAC-E2 placebo tablets and 1 moxifloxacin placebo capsule at Day -1.
  Once daily intake (orally) of 1 moxifloxacin placebo capsule at Day 14.
  Interventions: Drug: NOMAC-E2 (Org 10486-0 + Org 2317); Drug: Moxifloxacin placebo; Drug: NOMAC-E2 placebo
- Group C (Experimental): Once daily intake (orally) of 5 NOMAC-E2 (2.5/1.5 mg) tablets from Day 1 to Day 14.
  Once daily intake (orally) of 5 NOMAC-E2 placebo tablets and 1 moxifloxacin placebo capsule at Day -1.
  Once daily intake (orally) of 1 moxifloxacin placebo capsule at Day 14
  Interventions: Drug: NOMAC-E2 (Org 10486-0 + Org 2317); Drug: Moxifloxacin placebo; Drug: NOMAC-E2 placebo
- Group D (Placebo Comparator): Once daily intake (orally) of 5 NOMAC-E2 placebo tablets from Day -1 to Day 14.
  Once daily intake (orally) of 1 moxifloxacin placebo capsule at Days -1 and 14.
  Interventions: Drug: Moxifloxacin placebo; Drug: NOMAC-E2 placebo

INTERVENTIONS:
Drug: Moxifloxacin — Capsules containing 400 mg moxifloxacin, on Day 14 only
  Other Names: Avelox®
  Arms: Group A
Drug: NOMAC-E2 (Org 10486-0 + Org 2317) — Tablets containing 2.5 mg NOMAC and 1.5 mg E2, once daily dosing, orally taken. Daily dose either NOMAC-E2 2.5/1.5 mg or 12.5/7.5 mg.
  Arms: Group B; Group C
Drug: Moxifloxacin placebo — Moxifloxacin-placebo capsule taken orally, Day -1 and Day 14 only
Drug: NOMAC-E2 placebo — Tablets containing NOMAC-E2 placebo, once daily dosing, orally taken.

SUMMARY:
The trial is a single-center randomized, double-blind, double-dummy, placebo and positive controlled, parallel group clinical trial.

This trial investigated whether NOMAC-E2 (Org 10486 -0 + Org 2317), a new combined hormonal contraceptive, has potential to delay cardiac repolarization. The primary measure of cardiac repolarization in this trial is the Fridericia corrected QT interval (QTcF). QTcF represents the duration of ventricular depolarization and subsequent repolarization. A delay in cardiac repolarization creates an electrophysiological environment that favors the development of cardiac arrhythmias, most clearly torsade de pointes (TdP), but possibly other ventricular tachyarrhythmias.

The primary aim of this study is to investigate, if the administration of a therapeutic (2.5/1.5 mg) or supra-therapeutic (higher than required for treatment: 12.5/7.5 mg) dose of NOMAC-E2 administered over a period of 14 days will prolong the mean QTcF interval to values above the accepted threshold of regulatory concern.

In addition, a single dose of moxifloxacin will be administered in order to prove that sensitivity of the applied assay is sufficient to detect the prolongation of the QTcF-interval.

Secondary aims of this study are to evaluate the relation between concentrations of NOMAC (therapeutic and supra-therapeutic) after steady state has been reached in the subject's body, the time matched change in Estradiol E1 and E2 in relation to baseline and the QTcF intervals after multiple dose administration of NOMAC-E2.

Finally, the safety and tolerability of different treatments are investigated.

A total of 189 subjects will participate in this trial. The entire study duration is about 9 weeks with a 4-week screening period, 14-day treatment period and a follow-up period of about 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female (aged 18-50 years) with a body mass index (BMI) of 17 <= BMI <= 29 kg/m^2 at screening;
* Able and willing to use non-hormonal contraceptives during the trial from at least 2 weeks prior to Day 1 up to and including follow-up;
* Able and willing to sign the Informed Consent Form prior to screening evaluations;
* Subject is in a good age-appropriate healthy condition as established by medical history, physical examination, cardiac monitoring, electrocardiogram, results of biochemistry, hematology and urinalysis testing within 4 weeks prior to treatment as judged by the investigator;
* Normal 12-lead automatic ECG at screening and admission;
* Subject has a normal blood pressure at screening and admission;
* Subject smokes less than 5 cigarettes or equivalent per day and is capable of not smoking from 48 hours prior drug administration on Day -1 and Day 14 until the last ECG has been taken on respectively Day 1 and Day 15;
* Able to refrain from all use of (methyl)xanthines (e.g. coffee, tea, cola, chocolate) from 48 hours prior to drug administration on Day -1 and Day 14 until the last ECG has been taken on respectively Day 1 and Day 15;
* Able to refrain from alcohol containing beverages from 24 hours prior to drug administration on Day -1 and Day 14 until the last ECG has been taken on respectively Day 1 and Day 15;
* Able to refrain from all use of grapefruit containing products from 14 days prior to first NOMAC-E2 dosing until the last ECG has been taken;
* Easy venous accessibility.

Exclusion Criteria:

* History of sensitivity/idiosyncrasy to the applied drugs or chemically related compounds or excipients which may be employed in the study or to any other unknown drug used in the past
* Use of any drug or substance within one week and hormonal contraception within 2 weeks prior to the first treatment day, except for paracetamol or topical medication without systemic exposure
* Present use or use during 2 months prior to the start of treatment of any drugs interfering with the trial medication;
* Clinically relevant history or presence of any medical disorder, potentially interfering with this trial (according to the investigator)
* Known or suspected pregnancy
* History of/or current abuse of drugs or alcohol or solvents, or positive drug or alcohol screen at screening and admission, as judged by the (sub-)investigator
* Positive test result on hepatitis B surface antigen, hepatitis C antibody, or HIV 1/2 serology
* Participation in an investigational drug trial within 90 days prior to treatment
* Donation of blood within 90 days prior to treatment
* Contraindications for contraceptive steroids
* Breastfeeding or within 2 months after stopping breastfeeding prior to the start of trial medication.
* Present use or use within one month prior to treatment or within 10 half-lives in case the half-life > 3 days of any agent that is known to prolong the QT/QTc interval
* History of/or current risk factors for Torsade de Pointes (TdP) or life-threatening ventricular arrhythmia (e.g. heart failure, hypokaliemia, hypomagnesaemia, hypocalcaemia, family history of long or short QT syndrome, loss of consciousness)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2008-05; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Investigate whether once daily multiple therapeutic and supra-therapeutic doses of NOMAC-E2 prolong the mean QTcF interval at steady state to the threshold of regulatory concern compared to placebo | 16 days
Establish assay sensitivity after single dose of 400 mg moxifloxacin | 16 days

SECONDARY OUTCOMES:
evaluate the relation between steady state concentrations of NOMAC, time matched change from baseline in E1 and E2 and the QTcF intervals after multiple dosing of NOMAC-E2 | 16 days
Investigate safety and tolerability of the various treatments | 64 days

REFERENCES:
- [Derived] de Kam PJ, van Kuijk J, Lillin O, Post T, Thomsen T. The effect of therapeutic and supratherapeutic oral doses of nomegestrol acetate (NOMAC)/17beta-estradiol (E2) on QTcF intervals in healthy women: results from a randomized, double-blind, placebo- and positive-controlled trial. Clin Drug Investig. 2014 Jun;34(6):413-20. doi: 10.1007/s40261-014-0190-5. PMID 24777591